CLINICAL TRIAL: NCT02555865
Title: Aetiology of Children With Bronchiectasis in China--A Multicenter Retrospective Study
Brief Title: Aetiology of Children With Bronchiectasis in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Wuhan women and children's health care center (Unknown); Children's Hospital of Chongqing Medical University (Other); Yuying Children's Hospital of Wenzhou Medical University (Other); Changchun Children's Hospital (Other); Shenzhen Children's Hospital (Other Government); Jiangxi Province Children's Hospital (Other); Shanghai Children's Medical Center (Other); First Affiliated Hospital of Guangxi Medical University (Other); Tianjin Children's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department, Beijing Children's Hospital
Other Study IDs: BCHlung002
Record Dates: First submitted 2015-09-14; First posted 2015-09-22 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Bronchiectasis
Keywords: etiology; children
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This multicenter retrospective observation study is designed to investigate the etiology of children with bronchiectasis by review the medical records.

DETAILED DESCRIPTION:
This study is divided into two parts. Part I. Retrospective review the 10 years medical records of the children with bronchiectasis from every center, and investigate the etiology of the cases by the standard diagnostic process. Part II. All new cases of bronchiectasis which was confirmed diagnosed at every center from the beginning of the study are made the investigation of the etiology by the standard diagnostic process.

ELIGIBILITY:
Inclusion Criteria:A included patient must be coincident at least one point of the four items of HRCT manifestations.

* Internal bronchial diameter greater than the accompanying pulmonary artery.
* lack of bronchial tapering
* bronchi visible in the peripheral 1cm of lung
* bronchial diameter greater than adjacent segmental bronchi

Exclusion Criteria:Subject will be excluded if she or he has one of the following

* It is unable to provide complete medical records or the current condition can not accept the diagnosis process
* It does not agree to participate in the test

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as bronchiectasis at the certain hospitals (sponsor and collaborators)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with differential causes of bronchiectasis by reviewing the medical records or undergoing the standard diagnostic process | 48 months
  The cause of each paticipant with bronchiectasis will be recorded, for example post infection, PCD, PID, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD,PhD, Study Director — Beijing Children's Hospital of Capital Medical University, China; Baoping Xu, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China; Xiaoxia Peng, MD,PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China
Locations (1):
- Beijing Children'S Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Barker AF. Bronchiectasis. N Engl J Med. 2002 May 2;346(18):1383-93. doi: 10.1056/NEJMra012519. No abstract available. PMID 11986413
- [Background] Amorim A, Gracia Roldan J. Bronchiectasis: do we need aetiological investigation? Rev Port Pneumol. 2011 Jan-Feb;17(1):32-40. English, Portuguese. PMID 21251482
- [Background] Gaillard EA, Carty H, Heaf D, Smyth RL. Reversible bronchial dilatation in children: comparison of serial high-resolution computer tomography scans of the lungs. Eur J Radiol. 2003 Sep;47(3):215-20. doi: 10.1016/s0720-048x(02)00122-5. PMID 12927665
- [Background] Eastham KM, Fall AJ, Mitchell L, Spencer DA. The need to redefine non-cystic fibrosis bronchiectasis in childhood. Thorax. 2004 Apr;59(4):324-7. doi: 10.1136/thx.2003.011577. PMID 15047953
- [Background] Brower KS, Del Vecchio MT, Aronoff SC. The etiologies of non-CF bronchiectasis in childhood: a systematic review of 989 subjects. BMC Pediatr. 2014 Dec 10;14:4. doi: 10.1186/s12887-014-0299-y. PMID 25492164
- [Background] LIU Xiu-yun, JIANG Zai-fang. The etiology of ninety-one children with bronchiecatsis. J Clin Pediatr, 2011, 29(2):127-129.
- [Background] CHEN Jun, DUO Li-kun, WANG Xiao-feng. Clinical analysis of 22 children with bronchiectasis. J Clin Pediatr, 2012, 30(1):51-54.
- [Background] WANG Hao，XU Bao-ping，LIU Xiu-yun，HU Ying-hui，REN Yi-xin，SHEN Kun-ling. Clinical characteristics and follow-up of bronchiectasis in children. Chinese Journal of Practical Pediatrics, 2014;29 (12):936-939.